CLINICAL TRIAL: NCT05886803
Title: Prediction of the Spontaneous Breathing Test Success Using Biosignal and Biomarker in Critical Care Unit by a Machine Learning Approach
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Rea01
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Weaning From Mechanical Ventilation in Care Unit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous Breathing Test: The first group will be composed only by patients admitted in intensive care/critical care for ventilation support, and who successed the spontaneous breathing test.
  Interventions: Other: Spontaneous ventilation test
- Non Spontaneous Breathing Test: The second group will be composed only by patients admitted in intensive care/critical care for ventilation support, and who failed the spontaneous breathing test.
  Interventions: Other: Spontaneous ventilation test

INTERVENTIONS:
Other: Spontaneous ventilation test — The purpose is to mimic ventilation conditions after extubation and thus to help the clinician predict the outcome of an extubation decision.

SUMMARY:
Context:

Several authors have been interested in applying Artificial Intelligence (AI) to medicine, using various Machine Learning (ML) techniques: managing septic shock, predicting renal failure... [1, 2] AI has an important place in decision support for clinicians [3]. The weaning period is a really important time in the management of a patient on mechanical ventilation and can take up to half of the time spent in intensive care unit. The first weaning attempt is unsuccessful in 20% of patients However, mortality can be as high as 38% in patients with the most difficult weaning [4]. Only a few studies have looked at the application of machine learning in this area, and only one has looked at the use of biosignals (cardiac rate, ECG, ventilatory parameters…) [5-7]. To improve morbidity, mortality and reduce length of stay, it is essential to be able to predict the success of the spontaneous breathing test and extubation.

Investigators propose to develop a predictive algorithm for the success of a ventilatory weaning test based on biosignal records and others features.

Methods:

It is a critical care, oligo-centric and retrospective study the investigators included biosignal variables extracted from the electronic medical record, such as respiratory (RR, minute volume...), cardiac (systolic pressure, heart rate...), ventilator parameters and other discrete variables (age, comorbidity...). Most biosignal variables are minute-by-minute records. Recording starts 48 hours before the test and stops at the start of the weaning test. The investigators extracted features from these records, combined them with other biomarkers, and applied several machine learning algorithms: Logistic Regression, Random Forest Classifier, Support Vector Classifier (SVC), XGBoost, and Light Gradient Boosting Method (LGBM)…

ELIGIBILITY:
Inclusion Criteria:

* Computerized health report (CHR)
* Spontaneous breathing test should have been performed

Exclusion Criteria:

* Spontaneous breathing test has not been performed,
* Biosignal (cardiac, respiratory) are not registered in the CHR
* Patient died before the spontaneous breathing test
* Opposition to the study has been expressed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient admited in Intensive Care/Critical Care who needed ventilatory support, whatever the etiology requiring it.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of the spontaneous breathing test outcome. | 2 years
  Two modalities of test are performed in clinical : either a T-tube test or a spontaneous ventilation test at low level of Inspiratory Support and PEEP (7AI 4PEEP, 7Ai 0PEEP).
  A successful weaning test is defined by the absence of the following criteria at the end of the test: (i) increase in respiratory rate > 35cpm, (ii) SpO2 <90%, (iii) change of more than 20% in heart rate or blood pressure, (iv) modification of consciousness.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No